CLINICAL TRIAL: NCT01020461
Title: Evaluation of Accuvein for Blood Sampling and for Intravenous Catheter Placement in Adult Patients
Brief Title: Evaluation of Accuvein in Adult Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Arm "placement periph iv cath" COMPLETED - Arm "blood sampling" : study will not be performed because of the results of the arm "placement periph. iv cath"
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/43
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venous blood sampling (Experimental): To use Accuvein to improve the effectiveness of venous blood sampling
  Interventions: Device: Accuvein
- Peripheral IV catheter placement (Experimental): To use Accuvein to improve the effectiveness of placing peripheral IV catheter
  Interventions: Device: Accuvein

INTERVENTIONS:
Device: Accuvein — Accuvein will be used to facilitate venous blood sampling
  Arms: Venous blood sampling
Device: Accuvein — Accuvein will be used to facilitate peripheral IV catheter placement
  Arms: Peripheral IV catheter placement

SUMMARY:
The objective of this study is to evaluate the effectiveness of Accuvein to facilitate venous blood sampling and placement of peripheral intravenous catheters in adults. This clinical protocol is designed to determine whether using Accuvein increases the ease and efficiency of venous cannulation (as perceived by the operator), decreases the time to effective cannulation, decreases the number of sticks, and decreases the patient's perception of the pain.

ELIGIBILITY:
Inclusion Criteria:

* adults requiring a venous blood sampling or the placement of a venous peripheral catheter

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2010-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time to successful blood sampling or to successful placement of IV catheter | one hour

SECONDARY OUTCOMES:
Number of attempts required | Immediately after attempts
Pain | Immediately after attempts
Increases in the ease and efficiency of venous cannulation perceived by the operator) | Immediately after attempts

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Hôpital Foch, Suresnes, France, France

REFERENCES:
- [Derived] Aulagnier J, Hoc C, Mathieu E, Dreyfus JF, Fischler M, Le Guen M. Efficacy of AccuVein to facilitate peripheral intravenous placement in adults presenting to an emergency department: a randomized clinical trial. Acad Emerg Med. 2014 Aug;21(8):858-63. doi: 10.1111/acem.12437. PMID 25176152